CLINICAL TRIAL: NCT00402896
Title: Treatment of Malignant Pleural Effusion With ZD6474, a Novel Vascular Endothelial Growth Factor Receptor (VEGFR) and Epidermal Growth Factor Receptor (EGFR) Tyrosine Kinase Inhibitor
Brief Title: Malignant Pleural Effusion With ZD6474
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow Accrual
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2005-0929; NCI-2012-02082 (Registry Identifier: NCI CTRP); W81XWH-05-2-0027 (Other: DOD)
Record Dates: First submitted 2006-11-20; First posted 2006-11-22 (Estimated); Results first posted 2016-03-09 (Estimated); Last update posted 2016-03-09 (Estimated); Status verified 2016-02

CONDITIONS: Lung Cancer; Pleural Effusion
Keywords: Lung Cancer; Non-Small Cell Lung Cancer; Pleural Effusion; Indwelling Intrapleural Denver Catheter; ZD6474; Vascular Endothelial Growth Factor Receptor; VEGFR; Epidermal Growth factor Receptor; EGFR; Tyrosine Kinase Inhibitor
MeSH Terms: conditions — Lung Neoplasms; Pleural Effusion; Carcinoma, Non-Small-Cell Lung | interventions — vandetanib; Receptors, Vascular Endothelial Growth Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ZD6474 (Experimental): 300 mg/day orally for 10 weeks.
  Interventions: Drug: ZD6474

INTERVENTIONS:
Drug: ZD6474 — 300 mg/day orally for 10 weeks.
  Other Names: Vascular Endothelial Growth Factor Receptor; Epidermal Growth Factor Receptor Tyrosine Kinase Inhibitor

SUMMARY:
The goal of this clinical research study is to learn the effect of ZD6474 on the amount of time between placement of an indwelling pleural catheter and the catheter's removal in patients with malignant pleural effusion.

This study will also look at the effect that ZD6474 has on tumor cells, biological characteristics of cells in the body, rate of fluid build-up around the lungs, tumor size, and thickness of blood vessels. The effect that this drug has on quality of life and shortness of breath will also be examined.

DETAILED DESCRIPTION:
ZD6474 is an investigational drug that has not yet received approval from the FDA. ZD6474 is designed to limit VEGF. Vascular endothelial growth factor (VEGF) is considered to play a key role in the development of pleural effusion. Pleural effusion is an abnormal collection of pleural fluid in the pleural lining surrounding the lungs. The pleural lining is the thin covering that protects and cushions the lungs. It is made up of two layers of tissue that are separated by a small amount of fluid.

ZD6474 has shown promising activity against a number of cancers in laboratory tests in animals with cancer and in some early clinical trials in patients with non-small cell lung cancer (NSCLC). ZD6474 has also demonstrated significant reduction in pleural effusion in association with VEGF inhibition of tumor cells in mice with lung tumors and pleural effusion. It is hoped that ZD6474 will decrease the amount of pleural effusion that occurs in NSCLC patients. In addition, ZD6474 is thought to block the formation of new blood vessels, which may limit new blood vessel growth in the tumor and "starve" the tumor.

Before you can start treatment on this study, you will have "screening tests." These tests will help the doctor decide if you are eligible to take part in this study. You will have a complete physical exam, including measurement of vital signs (blood pressure, heart rate, temperature, and breathing rate), height, and weight. You will be asked questions about your ability to perform daily activities (performance status evaluation). You will have blood (about 2-3 teaspoons) drawn for routine tests. You may have up to 3 electrocardiograms (ECG --a test that measures the electrical activity of the heart). You will also have a chest x-ray and computed tomography (CT) scans of your chest to measure the status of the disease. You will be asked to fill out 2 questionnaires about the quality of your life and shortness of breath. The questionnaires will take about 10-15 minutes, total, to complete. Women who are able to have children must have a negative blood (about 1-2 teaspoons) pregnancy test.

If you are found to be eligible to participate in the study, you will have an indwelling intrapleural catheter placed. You will have to sign a separate consent document before placement of an indwelling intrapleural catheter can be performed. The pleural fluid will be collected at each clinic visit. The fluid will be saved and analyzed to answer research questions that are part of this study. You will also need to drain your pleural fluid everyday. The research nurse will provide you with instructions on how to drain your daily pleural fluid and a patient "diary" to take home to record the amount of fluid drained every day. The study doctor or research nurse will review the diary at each clinic visit.

After placement of the intrapleural catheter (Day 1), you will receive treatment with ZD6474. Treatment on this study is for 10 weeks. You will take a ZD6474 tablet by mouth each morning. The tablet should not be chewed, crushed, or divided, and should be taken with 8 ounces of water. You should take the tablet at about the same time every day.

During your participation on this study, you will have a physical exam, routine blood tests and chest x-ray at Weeks 2, 6, and 10. At Weeks 6 and 10, you will also have a CT scan. You will have an ECG at Weeks 1, 2, 4, and 8. Your doctor may decide to have additional ECGs to monitor your condition or if you experience a heart rate of less than 50 at any time during study participation. You will also be asked to complete 2 questionnaires about the quality of your life and any shortness of breath you are experiencing. You will complete these questionnaires at home and return them to the research staff at each clinic visit. You will be asked to record your weekly blood pressure for the first 6 weeks of study treatment. The study doctor or research nurse will review the log at each clinic visit.

If you are benefitting from the study treatment and your doctor feels that it is your best interest, you may continue to receive the study drug longer than 10 weeks. During your participation in this extended treatment phase, every 4 weeks you will have a physical exam and your performance status will be evaluated. You will have blood (about 2-3 teaspoons) drawn for routine tests. Every 4 weeks, you will have ECGs performed. You will also have a chest x-ray and computed tomography (CT) scans of your chest to measure the status of the disease every 8 weeks. Your study drug will continue to be provided to you.

You may be taken off study early if you have intolerable side effects or the disease gets worse.

This is an investigational study. ZD6474, the investigational drug to be used in this study, is not approved by the FDA for commercial use; however, the FDA has permitted its use in this research study. Up to 25 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with pleural effusion requiring placement of an indwelling intrapleural denver catheter for recurrent symptomatic malignant pleural effusion
2. Pathologic documentation of NSCLC
3. Performance status 0 to 2 (Eastern Cooperative Oncology Group (ECOG) scale)
4. International Normalized Ratio (INR) </= 2.5
5. Signed informed consent prior to any study related procedures
6. Subject must be female or male age 18 years or over

Exclusion Criteria:

1. Chemotherapy or other anticancer therapy in the 3 weeks prior to study. Palliative radiotherapy will be allowed to extra thoracic sites 2 weeks prior to study
2. No other prior malignancy is allowed except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or other cancer from which the patient has been disease-free for at least two years
3. Laboratory results sustained at:Neutrophils less than 1.5x10^9/L or platelets less than 100x10^9/L; Serum bilirubin >1.5 x the upper limit of reference range (ULRR);Serum creatinine>1.5xULRR or CrCl </=30 mL/minute(calculated by Cockcroft-Gault formula). Potassium,<4.0 mmol despite supplementation;serum calcium (ionized or adjusted for albumin),or magnesium out of normal range despite supplementation;Alanine aminotransferase(ALT)or aspartate aminotransferase(AST) > 2.5 x ULRR or alkaline phosphatase(ALP)> 2.5 x ULRR,or > 5 x ULRR if judged by the investigator to be related to liver metastases
4. Serious underlying medical condition that would impair the ability of the patient to receive protocol treatment, specifically cardiac diseases, uncontrolled hypertension or renal diseases
5. Diagnosis of post-obstructive pneumonia or other serious infection in the 14 days prior to registration
6. Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule
7. Evidence of severe or uncontrolled systemic disease or any concurrent condition which in the Investigator's opinion makes it undesirable for the patient to participate in the trial or which would jeopardize compliance with the protocol
8. Clinically significant cardiovascular event such as Myocardial infarction; New York Heart Association (NYHA) classification of heart disease >/=2 within 3 months before entry; or presence of cardiac disease that in the opinion of the Investigator increase the risk of ventricular arrhythmia
9. History of arrhythmia (multifocal premature ventricular contractions (PVCs), bigeminy, trigeminy, ventricular tachycardia, or uncontrolled atrial fibrillation) which is symptomatic or requires treatment (CTCAE grade 3) or asymptomatic sustained ventricular tachycardia. Atrial fibrillation, controlled on medication is not excluded
10. Previous history of corrected QT interval (QTc) prolongation with other medication that required discontinuation of that medication
11. Congenital long QT syndrome or 1st degree relative with unexplained sudden death under 40 years of age
12. QTc with Bazett's correction that is unmeasurable, or >/=480 msec on screening ECG. If a patient has QTc >/=480 msec on screening ECG, the screen ECG may be repeated twice (at least 24 hours apart). The average QTc from the three screening ECGs must be <480 msec in order for the patient to be eligible for the study). Patients who are receiving a drug that has a risk of QTc prolongation are excluded if QTc is >/= 460 msec
13. Any concomitant medication that may cause QTc prolongation or induce Torsades de Pointes
14. Hypertension not controlled by medical therapy (systolic blood pressure greater than 160 mm Hg or diastolic blood pressure greater than 100 mm Hg)
15. Women who are currently pregnant or breast feeding
16. Participation in a clinical trial of any investigational agents within 30 days prior to commencing study treatment
17. In 2nd line or later, the last dose of prior chemotherapy is discontinued less than 3 weeks before the start of study therapy
18. In 2nd line or later, the last radiation therapy discontinued less than 2 weeks before the start of study therapy except palliative radiotherapy
19. If it is in 2nd line or later, any unresolved toxicity greater than CTC grade 1 from previous anti-cancer therapy
20. Previous enrollment or randomization of treatment in the present study
21. Patients with pre-existing placement of intrapleural catheter
22. Presence of left bundle branch block (LBBB.)
23. Major surgery within 4 weeks, or incompletely healed surgical incision before starting study therapy
24. Patients may not have a history of a bleeding diathesis
25. Currently active diarrhea that may affect the ability of the patient to absorb the ZD6474 or tolerate diarrhea
26. Concomitant medications that are potent inducers (rifampicin, rifabutin, phenytoin, carbamazepine, phenobarbital and St. John's Wort) of CYP3A4 function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2006-10; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Jimenez, M.D., Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Massarelli E, Onn A, Marom EM, Alden CM, Liu DD, Tran HT, Mino B, Wistuba II, Faiz SA, Bashoura L, Eapen GA, Morice RC, Jack Lee J, Hong WK, Herbst RS, Jimenez CA. Vandetanib and indwelling pleural catheter for non-small-cell lung cancer with recurrent malignant pleural effusion. Clin Lung Cancer. 2014 Sep;15(5):379-86. doi: 10.1016/j.cllc.2014.04.002. Epub 2014 May 14. PMID 24913066
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: October 2006 to July 2010 at UT MD Anderson Cancer Center included NSCLC participants diagnosed with proven metastatic disease to the pleural space by pleural fluid cytology or pleural biopsy and required IPC placement because of symptomatic recurrent pleural effusions between May 2007 and February 2010.
Pre-assignment Details: The clinical trial was terminated before reaching the target patient accrual due to ZD6474 unavailability and of the 28 enrolled but only 20 received treatment. Slow accrual was a contributing factor to early termination.
Period: Overall Study
Arm/Group | ZD6474
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | ZD6474
Number analyzed (Participants) | 20
Age, Continuous [Median (Full Range); unit: years] | 72 [46 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 11
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Median Time to Pleurodesis
Description: Time to pleurodesis from initiation of treatment to catheter removal as measure of pleural effusion Improvement (amount of pleural fluid drainage) where objective was to examine whether ZD6474 would help participants to improve the condition of pleural effusion, and thus remove the catheter earlier. Cox model analysis applied to examine the effect of covariates on the time to catheter removal.
Time Frame: Time from initiation of treatment and catheter insertion up to a maximum of 10 weeks
Population: Twenty eligible participants were analyzed for the primary outcome in the trial, eleven completed 10 weeks of treatment. All twenty participants completed the study.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | ZD6474
Number analyzed (Participants) | 20
Days | 35 [15 to NA] — Distributional assumptions were not available making it not possible to obtain an exact 95% confidence interval for the median.

ADVERSE EVENTS:
Time Frame: Adverse event collection for 10 week treatment period. Collection period: May 2007 to February 2010.
Arm/Group | ZD6474
Serious Adverse Events (participants affected / at risk) | 12/20
Other Adverse Events (participants affected / at risk) | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ZD6474 (N=20)
CNS Ischemia (Nervous system disorders) | 1 (1) — Transient Ischemic Attack
Creatinine (Renal and urinary disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pain (General disorders) | 1 (1)
Motor Neuropathy (Nervous system disorders) | 1 (1)
Dehydration (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Weight Loss (General disorders) | 1 (1)
Left Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
R. Pneumothorax (Infections and infestations) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ZD6474 (N=20)
Anemia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 2 — partial thromboplastin time (PTT)
Prolonged PTT (Blood and lymphatic system disorders) | 1
Fatigue (General disorders) | 7
Weight loss (General disorders) | 5
Anorexia (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 12
Constipation (Gastrointestinal disorders) | 1
Xerostomia (Gastrointestinal disorders) | 2
Abdominal Distension/bloating (Gastrointestinal disorders) | 1
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Prolonged QTc (Cardiac disorders) | 5
Cardiac arrhythmia (Cardiac disorders) | 3
Palpitations (Cardiac disorders) | 1
Hypertension (Cardiac disorders) | 1
Premature ventricular contractions (Cardiac disorders) | 1
Acne (Skin and subcutaneous tissue disorders) | 2
Dry skin (Skin and subcutaneous tissue disorders) | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 4
Rash/desquamation (Skin and subcutaneous tissue disorders) | 4
Sweating (General disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Infection with normal ANC (Infections and infestations) | 1
Hypomagnesemia (Blood and lymphatic system disorders) | 5
Hypokalemia (Blood and lymphatic system disorders) | 4
Hyponatremia (Blood and lymphatic system disorders) | 1
Hypophosphatemia (Blood and lymphatic system disorders) | 3
Hyperkalemia (Blood and lymphatic system disorders) | 1
Dizziness (Nervous system disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes